CLINICAL TRIAL: NCT04344886
Title: Optimization and Individualization of Diagnostic Scintigraphy Protocol and Minimally Invasive Radio-guided Parathyroid Surgery Using Quantitative Analysis of Scintigraphy Results on Hybrid SPECT-CT Imaging
Brief Title: Optimization and Individualization of Diagnostic Scintigraphy Protocol and Minimally Invasive Radio-guided Parathyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-ENT-Parathyroid_adenoma
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Primary Hyperparathyroidism; Thyroid Disease; Parathyroid Diseases; Parathyroid Adenoma
Keywords: minimally-invasive radio-guided parathyroidectomy; in-vivo; ex-vivo; multi-phase SPECT/CT; individualized treatment
MeSH Terms: conditions — Hyperparathyroidism, Primary; Thyroid Diseases; Parathyroid Diseases; Parathyroid Neoplasms | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: The patients are randomized into two parallel study arms.
Masking Description: No masking is being used in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (dual-phase) SPECT/CT (Experimental): Adult patients with primary hyperparathyroidism undergoing conventional (dual-phase) SPECT/CT (after 10 and 150 minutes) and conventional minimally-invasive radio-guided parathyroidectomy in a time span 2-3 hours from radionuclide administration.
  Interventions: Procedure: Conventional (dual-phase) SPECT/CT; Procedure: Conventional minimally-invasive radio-guided parathyroidectomy
- Multi-phase SPECT/CT (Experimental): Adult patients with primary hyperparathyroidism undergoing multi-phase SPECT/CT (after 10, 90, 150, 210 minutes) and individualized minimally-invasive radio-guided parathyroidectomy performed in a recommended time span based on standardized uptake value calculation.
  Interventions: Procedure: Multi-phase SPECT/CT; Procedure: Individualised minimally-invasive radio-guided parathyroidectomy

INTERVENTIONS:
Procedure: Conventional (dual-phase) SPECT/CT — Conventional (dual-phase) SPECT/CT (after 10 and 150 minutes)
  Arms: Conventional (dual-phase) SPECT/CT
Procedure: Multi-phase SPECT/CT — Multi-phase SPECT/CT (after 10, 90, 150, 210 minutes)
  Arms: Multi-phase SPECT/CT
Procedure: Conventional minimally-invasive radio-guided parathyroidectomy — Conventional minimally invasive radio-guided parathyroidectomy in a time span of 2-3 hours from radionuclide administration
  Arms: Conventional (dual-phase) SPECT/CT
Procedure: Individualised minimally-invasive radio-guided parathyroidectomy — Individualized minimally-invasive radio-guided parathyroidectomy performed in a recommended time span based on standardized uptake value calculation.
  Arms: Multi-phase SPECT/CT

SUMMARY:
The radio-guided technique offers both help with in-vivo identification and ex-vivo confirmation of parathyroid adenoma. In-vivo accuracy is most important but its results are not satisfactory. The aim of this study was to evaluate if there is a beneficial effect of individualized timing of surgery using preoperative multi-phase 99mTc-MIBI single-photon emission computed tomography (SPECT)/CT on in-vivo characteristics of minimally invasive radio-guided parathyroidectomy.

DETAILED DESCRIPTION:
Despite the relatively accurate preoperative topographic information, minimally invasive parathyroid surgery can still be very challenging, especially in the case of small adenoma in ectopic localization. Radioguided technique offers both help with in-vivo identification and ex-vivo confirmation of adenoma. Excellent ex-vivo radio guidance results are referred. But, in-vivo accuracy is most important but its results are not satisfactory. The aim of this study was to evaluate if there is a beneficial effect of individualized timing of surgery using preoperative multi-phase 99mTc-MIBI single-photon emission computed tomography (SPECT)/CT on in-vivo characteristics of minimally invasive radio-guided parathyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* No history of thyroid or parathyroid surgery
* Diagnosis of primary hyperparathyroidism
* Indication for 99mTc-MIBI SPECT/CT examination

Exclusion Criteria:

* Minor patients
* Negative SPECT/CT findings
* Patients refusing surgery
* Previous combined surgery on the thyroid gland
* Patients in high risk of general anesthesia
* Patients who do not undergo surgery in the recommended time span

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Success of surgery (%) | 3 months
  Surgery was considered successful if there were lowering of parathyroid hormone serum level and calcemia to normal and histological confirmation of parathyroid gland adenoma/ hyperplasia.
In-vivo sensitivity (%) | 3 months
  Calculated from number of true positive, false positive, true negative and false negative cases identified by gamma probe during surgery. The parathyroid tissue was considered pathologic when the in-vivo radioactive counting was at least 1.15 times more than the background.
In-vivo specificity (%) | 3 months
  Calculated from number of true positive, false positive, true negative and false negative cases identified by gamma probe during surgery. The parathyroid tissue was considered pathologic when the in-vivo radioactive counting was at least 1.15 times more than the background.
In-vivo accuracy (%) | 3 months
  Calculated from number of true positive, false positive, true negative and false negative cases identified by gamma probe during surgery. The parathyroid tissue was considered pathologic when the in-vivo radioactive counting was at least 1.15 times more than the background.
Ex-vivo sensitivity (%) | 3 months
  Calculated from number of true positive, false positive, true negative and false negative cases identified by gamma probe during surgery. Radioactive ex-vivo counts in adenoma/ hyperplastic parathyroid gland greater than 20% of background was used as cutpoint for cure.
Ex-vivo specificity (%) | 3 months
  Calculated from number of true positive, false positive, true negative and false negative cases identified by gamma probe during surgery. Radioactive ex-vivo counts in adenoma/ hyperplastic parathyroid gland greater than 20% of background was used as cutpoint for cure.
Ex-vivo accuracy (%) | 3 months
  Calculated from number of true positive, false positive, true negative and false negative cases identified by gamma probe during surgery. Radioactive ex-vivo counts in adenoma/ hyperplastic parathyroid gland greater than 20% of background was used as cutpoint for cure.

SECONDARY OUTCOMES:
Operating time (minutes) | Duration of surgery
  The operating time will be measured and recorded.
Pathological parathyroid gland volume (ml) | Duration of surgery
  The pathological parathyroid gland volume in millilitres will be measured and recorded.
Pathological parathyroid gland localisation (ectopic x eutopic) | Duration of surgery
  The pathological parathyroid gland localisation (ectopic x eutopic) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimír Dedek, MD,PhD, Study Chair — University Hospital Ostrava; Martin Formánek, MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be made available to other researchers upon request.